CLINICAL TRIAL: NCT06758440
Title: Effectiveness of Hydroxyapatite Reinforced Chitosan Hydrogel in Modulation of Osseintegration Round Immediate Dental Implant Randomized Single Blind Control Study
Brief Title: Effectiveness of Hydroxyapatite Reinforced Chitosan Hydrogel in Modulation of Osseointegration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Tarek Abdelbarry, Lecturer of Oral and Maxillofacial Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Osseintegration
Record Dates: First submitted 2023-05-16; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2023-03

CONDITIONS: Osseointegration Failure of Dental Implant
MeSH Terms: interventions — Chitosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 10 patients injected by chitosan/ hydroxyapatite hydrogel in the extracted socket in a back fill injection manner prior to immediate implant placement and then covered with HemCon dental dressing Pro
  Interventions: Drug: chitosan
- Group B (Active Comparator): About 10 patients received dental immediate implant placement Spectra system
  Interventions: Drug: chitosan

INTERVENTIONS:
Drug: chitosan — Evaluate Effectiveness of hydroxyapatite reinforced chitosan hydrogel in modulation of osseintegration round immediate dental implant in a Randomized single blind control study
  Other Names: hydroxyapatite hydrogel

SUMMARY:
Dental implant treatments have now become indispensable in clinical dental practice. The survival rate exceeds 90%; Modern oral implantology uses different devices, in terms of size, shape, length, thickness and composition, from pure titanium to titanium-aluminum-vanadium alloys, due to their biocompatibility and high corrosion resistance

DETAILED DESCRIPTION:
Immediate implants placed in freshly extracted sockets are an alternative treatment for traditional dental implants reduces physiological resorption of alveolar ridge, provides fast and simple procedures , decreasing the number of dental appointments, shortening length of treatment time, lesser surgical intervention, and ideal axial orientation of the implant.

However, the biological response of tissues can be improved by different surface treatments that provide both bioactivity and osseointegration capacity. Many materials have been advocated for boosting up the bone regeneration.

Current trends are directed not only towards achieving optimal osseointegrative surfaces, but also towards antibacterial activity for prolonged periods of time, either by blocking microbial adhesion and preventing late infections.

Given their biocompatibility and biodegradability, natural polymers are widely used materials for bone grafting. Among them, chitosan, collagen, silk fibroin, gelatin, cellulose, alginate. Chitosan is an excellent candidate for bone reconstruction as it has antimicrobial properties, can generate porous structures suitable for cell growth and osteoconduction, and promotes osteoblast cell proliferation. Furthermore, its structure is similar to glycosaminoglycans, a component of the bone extracellular matrix.

Chitosan has been formulated in different systems for bone tissue engineering, including scaffolds, sponges, hydrogels, micro-nanospheres, and membranes, among others ; capable of accelerating the formation of new bone integrated into the host bone without causing adverse reactions .

A large number of studies on chitosan-based gel scaffolds for bone regeneration can be found in the literature. It is usual to develop systems that combine chitosan with other compounds as hydroxyapatite to improve properties such as osteoconductivity and mechanical properties and thus obtain materials that mimic natural bone as much as possible.

Hydrogels have also been studied for surgical applications. These systems consist of a liquid phase, which generally comprises 90% of the formulation, trapped in a solid phase that gives the gel its structure . This water content makes these systems highly biocompatible, and their soft consistency prevents damage to surrounding tissues. Chitosan hydrogels show similar mechanical properties to connective tissues, which favors tissue regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (class I category according to American society of anesthesiologists )
* Over 20 years and under 50 years of age
* Either gender
* Patients seeking extraction and placement of immediate dental implant for mandibular teeth.

Exclusion Criteria:

* Any acute infection in surgical sites
* Long term non-steroidal anti-inflammatory drug therapy
* Periodontal disease with bone loss
* Known allergy to any of the materials used in the study
* Patients with severely atrophic ridges requiring a staged grafting procedure
* Patients with significant medical condition
* Alcoholic individuals
* Patients on drugs that affect the central nervous systems
* Patients who reported the use of drugs that might interfere with pain sensitivity
* Pregnant and lactating

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of osseintegration | 6 months
  Early follow up was performed daily for appearing any complications pre-operative or post-operative.

SECONDARY OUTCOMES:
Radiographic assessment | 6 months
  Difference in bone density (in Hounsfield units) using CBC and marginal bone level in mm using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No